CLINICAL TRIAL: NCT00839995
Title: A Prospective Observational Study to Evaluate Perioperative Coagulation Profiles Using Rotational Thromboelastometry (ROTEM®) in Patients Undergoing Multi-level Spine Surgery
Brief Title: Use of ROTEM for Multi-level Spine Surgery
Acronym: ROTEM
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Hugh Hemmings, Vice Chair of Research, Weill Medical College of Cornell University
Other Study IDs: 0811010079
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-02

CONDITIONS: Coagulation
Keywords: To determine the efficacy of ROTEM on assessing coagulation profiles.
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — a small sample of blood will be obtained from a pre-existing arterial line.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing multi-level spine surgery

SUMMARY:
The purpose of this study is to obtain coagulation profiles of patients undergoing multi-level spine surgeries with ROTEM® and routine coagulation tests. The investigators will compare the data from ROTEM® and routine coagulation tests with each other and with blood loss and transfusion therapies used.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective open spine (cervical, thoracic, and/or lumbar) surgery with anticipated blood loss of > 1 L
* Males and females
* Age 18 to 100 years of age
* ASA physical status 1 to 3
* Arterial line indicated for the intraoperative management of the patient and in place prior to incision
* Informed consent obtained

Exclusion Criteria:

* Known pre-existing hemostatic abnormality
* Known clopidogrel use within 10 days prior to surgery
* Known warfarin use within 5 days prior to surgery
* Known pregnancy
* Has physical, mental, or medical conditions which, in the opinion of the Investigator, could compromise the subject's welfare, ability to communicate with the study staff, complete study activities, or would otherwise contraindicate study participation.
* Inclusion in another clinical research study
* An investigator of this study
* Subject's refusal or inability to agree to and sign the Informed Consent form in English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Large metropolitan hospital.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Coagulation profiles. | One measurement before surgery, one after surgery is completed, and one measurement at each i-stat or 10% total blood volume loss.

CONTACTS AND LOCATIONS:
Overall Officials: Hugh C Hemmings, M.D., Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Background] Mannucci PM, Levi M. Prevention and treatment of major blood loss. N Engl J Med. 2007 May 31;356(22):2301-11. doi: 10.1056/NEJMra067742. No abstract available. PMID 17538089
- [Background] Kozek-Langenecker S. Management of massive operative blood loss. Minerva Anestesiol. 2007 Jul-Aug;73(7-8):401-15. Epub 2007 Mar 27. PMID 17380100
- [Background] Ebinger T. Concerning Hanecke P, Klouche M: Thrombelastography Today: Practicability and Analytical Power. Transfus Med Hemother 2007;34:421-428. Transfus Med Hemother. 2008;35(4):324-326. doi: 10.1159/000143229. Epub 2008 Jul 21. No abstract available. PMID 21512650
- [Background] Hu SS. Blood loss in adult spinal surgery. Eur Spine J. 2004 Oct;13 Suppl 1(Suppl 1):S3-5. doi: 10.1007/s00586-004-0753-x. Epub 2004 Jun 10. PMID 15197630
- [Background] Luddington RJ. Thrombelastography/thromboelastometry. Clin Lab Haematol. 2005 Apr;27(2):81-90. doi: 10.1111/j.1365-2257.2005.00681.x. PMID 15784122
- [Background] Yuan S, Ferrell C, Chandler WL. Comparing the prothrombin time INR versus the APTT to evaluate the coagulopathy of acute trauma. Thromb Res. 2007;120(1):29-37. doi: 10.1016/j.thromres.2006.07.002. Epub 2006 Aug 2. PMID 16887171
- [Background] Ciavarella D, Reed RL, Counts RB, Baron L, Pavlin E, Heimbach DM, Carrico CJ. Clotting factor levels and the risk of diffuse microvascular bleeding in the massively transfused patient. Br J Haematol. 1987 Nov;67(3):365-8. doi: 10.1111/j.1365-2141.1987.tb02359.x. PMID 3689699
- [Background] Segal JB, Dzik WH; Transfusion Medicine/Hemostasis Clinical Trials Network. Paucity of studies to support that abnormal coagulation test results predict bleeding in the setting of invasive procedures: an evidence-based review. Transfusion. 2005 Sep;45(9):1413-25. doi: 10.1111/j.1537-2995.2005.00546.x. PMID 16131373
- [Background] Ganter MT, Hofer CK. Coagulation monitoring: current techniques and clinical use of viscoelastic point-of-care coagulation devices. Anesth Analg. 2008 May;106(5):1366-75. doi: 10.1213/ane.0b013e318168b367. PMID 18420846
- [Background] American Society of Anesthesiologists Task Force on Perioperative Blood Transfusion and Adjuvant Therapies. Practice guidelines for perioperative blood transfusion and adjuvant therapies: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Blood Transfusion and Adjuvant Therapies. Anesthesiology. 2006 Jul;105(1):198-208. doi: 10.1097/00000542-200607000-00030. No abstract available. PMID 16810012
- [Background] Spalding GJ, Hartrumpf M, Sierig T, Oesberg N, Kirschke CG, Albes JM. Cost reduction of perioperative coagulation management in cardiac surgery: value of "bedside" thrombelastography (ROTEM). Eur J Cardiothorac Surg. 2007 Jun;31(6):1052-7. doi: 10.1016/j.ejcts.2007.02.022. Epub 2007 Mar 29. PMID 17398108